CLINICAL TRIAL: NCT00226226
Title: Peripherally Inserted Central Catheter Placement by IV Team Nurses Using the Sonic Flashlight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0506042
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Catheterization

INTERVENTIONS:
Procedure: Peripherally Inserted Central Catheter Placement

SUMMARY:
The purpose of this study is to test whether peripherally inserted central catheters can be safely placed on patients by intravenous team nurses at the bedside.

DETAILED DESCRIPTION:
We have developed a new device for guiding invasive procedures with ultrasound (US), which we call the Sonic Flashlight (SF). We attach a half-silvered mirror and a small flat-panel monitor directly to an ultrasound transducer to project a virtual image of the US scan into its actual location within the patient. This permits the operator to guide a needle through the skin by aiming directly at the image, using natural hand-eye coordination rather than looking away from the patient at a conventional display. We believe the SF will increase accuracy, safety, and speed for a wide variety of invasive procedures and yield a faster learning of these procedures than conventional US displays.

The research proposed here would bring the application of guided needle insertion to its clinical implementation, specifically addressing the placement of the Peripherally Inserted Central Catheter (PICC) line. The PICC line is increasingly viewed as a safe alternative to direct central line placement in the jugular, subclavian, and femoral veins, while being easier to maintain than a peripheral intravenous line. This study will test the hypothesis that PICC lines can be placed by experienced intravenous (IV) team nurses using the SF for real-time US guidance.

Thirty nurse participants (ages 18-65) will be recruited from the IV team at UPMC Presbyterian Hospital to participate in the study. 200 patient subjects will be recruited from the adult (18 years and older) population of patients already scheduled to receive the PICC placement procedure; patients will have the lines placed by experienced IV team nurses using ultrasound guidance with either the SF or conventional ultrasound (CUS). Investigators will observe each procedure, using audio and video recording, ultrasound image data, and other characteristics of the procedure to monitor the success of each procedure. A set of feasibility trials will be conducted in the interventional radiology (IR) suite to assess the level of training the nurses have received prior to the start of the comparison trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Undergoing peripherally inserted central catheter placement as standard of care.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2006-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
PICC line successfully placed by intravenous team nurses using the Sonic Flashlight

SECONDARY OUTCOMES:
PICC line successfully placed by intravenous team nurses using conventional ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: George D Stetten, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States